CLINICAL TRIAL: NCT02554370
Title: Psychoeducational Programme for Patients With Parkinson's Disease Undergoing Subthalamic Deep Brain Stimulation
Brief Title: Psychoeducational Programme for PD Patients With STN-DBS
Acronym: PSYCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Marie-laure Welter, Medical Doctor, Groupe Hospitalier Pitie-Salpetriere
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2006-A00230-51
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational programme (Experimental): Psychoeducational programme
  Interventions: Behavioral: Psychoeducational programme
- Usual care (No Intervention): No psychoeducational programme

INTERVENTIONS:
Behavioral: Psychoeducational programme — 4 sessions of psychoeducation before and 3 after surgery for subthalamic deep brain stimulation
  Arms: Psychoeducational programme

SUMMARY:
Bilateral subthalamic deep-brain stimulation is a well-established therapeutic option to improve motor signs and reduce dopaminergic treatment and related motor complications in patients with severe forms of Parkinson's disease (PD). However, psychological disorders and socio-familial maladjustment are less clearly improved with subthalamic stimulation with an aggravation of the social adjustment described in about 1/3 of cases, with work disruption, divorce or familial conflict. The caregivers have also been reported to present negative well-being after surgery with an aggravation of the quality of life. In the present study, the investigators evaluate the effects of a perioperative psychoeducational programme to avoid postoperative socio-familial maladjustment in PD patients candidate for subthalamic stimulation, and their caregivers, in a randomized controlled study.

DETAILED DESCRIPTION:
After inclusion, patients (and their caregivers) are randomized into two groups stratified on their preoperative social adjustment scale couple domain score : usual treatment and psychoeducational programme or usual treatment alone (Figure). The psychoeducational programme focuses on 3 domains: 1) neurosurgical procedure and neurological outcome, 2) social life including work, social and familial relationship, 3) couple relationship. The programme consists of 7 sessions with 3 to 4 couples at the same session, except for the 'couple relationship' domain. Each domain is tackled in a two-way manner with information/education proved by the investigator and discussion of the patients' and caregivers' expectations during one session. The following session started with a 'Questions and Answers' on the previous domain and then information on another domain. Four sessions were carried out prior to surgery and 3 after.

ELIGIBILITY:
Inclusion Criteria:

* Parkison's disease
* Patients candidate for STN DBS
* Caregiver agreeing to participate
* Signed informed consent

Exclusion Criteria:

* Contra-indication to STN-DBS
* No caregiver agreeing to participate
* Dementia
* Severe ongoing psychiatric disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Social adjustment scale | Change from baseline at 1 year after surgery

SECONDARY OUTCOMES:
Parkinson's disease Questionnaire PDQ-39 | Change from baseline at 1 and 2 years after surgery
  Quality of life
Anxiety scale (STAI) | Change from baseline at 1 and 2 years after surgery
  STAI
Mattis dementia rating scale | Change from baseline at 1 and 2 years after surgery
  mattis dementia rating scale
Parkinsonian disability (Unified Parkinson's Disease Rating Scale) | Change from baseline at 1 and 2 years after surgery
  Unified Parkinson's Disease Rating Scale
Dopaminergic treatment dosage (mg/day) | Change from baseline at 1 and 2 years after surgery
  Daily dosage of dopaminergic agents
Social adjustment scale | Change from baseline at 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Vacher, Study Chair — APHP
Locations (1):
- Centre d'Investigation Clinique GHPS, Paris, Paris, France